CLINICAL TRIAL: NCT02527772
Title: Liposomal Doxorubicin(LD) Plus Gemcitabine Versus Oxaliplatin Plus Fluorouracil/Leucovorin(FOLFOX4) As Palliative Chemotherapy in Patients With Advanced Hepatocellular Carcinoma(HCC)
Brief Title: Liposomal Doxorubicin Plus Gemcitabine Versus Oxaliplatin Plus Fluorouracil/Leucovorin for Hepatocellular Carcinoma
Acronym: LD-FOX4/HCC
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: It doesn't meet the requirements of randomized trials
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Liao, Affiliated Tumor Hospital, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LD-FOX4/HCC
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — liposomal doxorubicin; Gemcitabine; Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Doxorubicin+Gemcitabine (Experimental): Gemcitabine 1000mg/m2,d1,8;Liposomal Doxorubicin 30mg/m2,d1.q4w
  Interventions: Drug: Liposomal Doxorubicin+Gemcitabine
- FOLFOX4 (Active Comparator): Oxaliplatin 85 mg/m2 intravenously on day 1; Leucovorin 200 mg/m2 IV(in vein) from hour 0 to 2 on days 1 and 2; and Fluorouracil 400 mg/m2 IV bolus at hour 2, then 600mg/m2 over 22 hours on days 1 and 2, once every 2 weeks
  Interventions: Drug: FOLFOX4

INTERVENTIONS:
Drug: Liposomal Doxorubicin+Gemcitabine — Gemcitabine 1000mg/m2,d1,8,iv; Liposomal Doxorubicin 30mg/m2,d1,iv.q4w of each 28 day cycle. 6 of Cycles: until progression or unacceptable toxicity develops or Progressive Disease.
  Other Names: Liposomal Doxorubicin plus Gemcitabine
  Arms: Liposomal Doxorubicin+Gemcitabine
Drug: FOLFOX4 — Oxaliplatin 85 mg/m2 intravenously on day 1; Leucovorin 200 mg/m2 IV(in vein) from hour 0 to 2 on days 1 and 2; and Fluorouracil 400 mg/m2 IV bolus at hour 2, then 600mg/m2 over 22 hours on days 1 and 2, once every 2 weeks until progression or unacceptable toxicity develops or Progressive Disease.
  Other Names: Oxaliplatin plus Fluorouracil/Leucovorin
  Arms: FOLFOX4

SUMMARY:
The purpose of this study is to determine that Liposomal Doxorubicin(LD) plus Gemcitabine(GEM) is superior to Oxaliplatin（OXA） Plus Fluorouracil/Leucovorin(FOLFOX4) in prolonging progression-free survival（PFS） in patients with Advanced Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were age 18 to 75 years;
* The patients had histologically, cytologically,or clinically diagnosed unresectable HCC;and were ineligible for local invasive treatment. Clinically diagnosed patients had to have: (1) evidence of HBV or HCV with hepatic cirrhosis; (2) a-fetoprotein levels 400g/L; and (3) morphologic evidence of hypervascular liver tumor. Patients had to have at least one measurable lesion according to RECIST (version 1.0; ≥2 cm on computed tomography [CT]; 1 cm on spiral CT or magnetic resonance imaging). Lesions that had undergone previous interventional or local therapy were not considered measurable lesions.
* ECOG score≤2;
* life expectancy 3 months;
* Barcelona Clinic liver cancer (BCLC) stage B or C disease;
* Child-Pugh stage A or B disease;
* Adequate organ and marrow function, with neutrophil count≥1.5X10e9/L, platelet count≥75×10e9/L, AST or ALT﹤2.5×upper limit of normal (ULN), total bilirubin <1.5×ULN, international normalized ratio <1.5;normal baseline left ventricular ejection fraction_lower limit of normal for the institution. Patients with AST and ALT< 5 ×ULN could be recruited if total bilirubin was in the normal range.
* Patients had to provide signed informed consent to participate.

Exclusion Criteria:

* documented allergy to platinum compounds or other study drugs; any previous OXA or DOX treatment, except adjuvant treatment ﹥12 months before random assignment;
* Previous liver transplantation;
* concomitant use of any other anticancer therapy, including interferon alfa and herbal medicine approved by the local authority to be used as anticancer medicine (except palliative radiotherapy to a nontarget lesion);
* CNS metastasis;
* Other serious illness or medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free-Survival | 6 months

SECONDARY OUTCOMES:
Objective response rate | 3 months
Overall survival | 6 months and 12 months
Disease control rate | 3 months
Time-to-Progression | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: lequn Li, MD, Study Director — GXMU

REFERENCES:
- [Result] Lombardi G, Zustovich F, Farinati F, Cillo U, Vitale A, Zanus G, Donach M, Farina M, Zovato S, Pastorelli D. Pegylated liposomal doxorubicin and gemcitabine in patients with advanced hepatocellular carcinoma: results of a phase 2 study. Cancer. 2011 Jan 1;117(1):125-33. doi: 10.1002/cncr.25578. Epub 2010 Aug 31. PMID 21058409
- [Result] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077